CLINICAL TRIAL: NCT04255134
Title: Comparison of Abatacept With Tumor Necrosis Factor Inhibitors in the Treatment of Rheumatoid Arthritis Pain: A Phase IV Trial
Brief Title: Biologics for Rheumatoid Arthritis Pain (BIORA-PAIN)
Acronym: BIORA-PAIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019.0146
Record Dates: First submitted 2019-11-14; First posted 2020-02-05 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept; Adalimumab

STUDY DESIGN:
Masking Description: This is a randomized, open label trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abatacept (Experimental): Drug administered to participants with active rheumatoid arthritis
  Interventions: Drug: Abatacept Injection
- Adalimumab (Active Comparator): Comparator drug administered to participants with active rheumatoid arthritis
  Interventions: Drug: Adalimumab Injection

INTERVENTIONS:
Drug: Abatacept Injection — Subjects will be randomized to treatment with either abatacept or adalimumab
  Other Names: Orencia
  Arms: Abatacept
Drug: Adalimumab Injection — Subjects will be randomized to treatment with either abatacept or adalimumab
  Other Names: Humira
  Arms: Adalimumab

SUMMARY:
It is increasingly recognized that although suppression of inflammation is a treatment goal in rheumatoid arthritis, many people who have control of their inflammation continue to experience pain. A number of studies have recently shown that by measuring further characteristics of pain in rheumatoid arthritis, e.g. neuropathic pain, quantitative sensory testing, compared with objective measures of inflammation, it is possible to acquire more detailed information about the level of pain in relation to inflammation that a patient with rheumatoid arthritis is experiencing, which could assist in developing their care.

In this study, the investigators will explore validated endpoints for pain including the Visual Analogue Scale for pain, neuropathic pain scores and quantitative sensory testing for pain.

The investigators will evaluate in a population-based study, the pain profile using the Visual Analog Scale (VAS), neuropathic pain assessment, quantitative sensory testing (QST) by pain pressure thresholds (PPT) in comparison to markers of inflammation in order to assess the difference in pain outcomes between baseline pre- and post- treatment in a population of participants with active Rheumatoid Arthritis treated with abatacept and Tumor Necrosis Factor (TNF) inhibitors respectively. All measures will be conducted systematically in the abatacept and TNF inhibitor groups pre- and post-treatment with respective biologic agents. Participants with active Rheumatoid Arthritis who may be eligible for biologic treatment will be screened for enrolment into the study.

DETAILED DESCRIPTION:
Primary objective To examine: Pain characteristics in participants with active rheumatoid arthritis receiving abatacept biologic therapy versus TNF inhibitor therapy in the form of adalimumab.

To establish if there are differences in pain outcomes by patient reported scores, objective measures of pain using quantitative sensory testing and inflammatory markers in participants receiving biologic therapies for rheumatoid arthritis.

Population: The population being assessed in this study are participants with active rheumatoid arthritis with a disease activity score of greater than 5.1.

Intervention: Subjects will be randomized to treatment with abatacept or adalimumab for active rheumatoid arthritis

Comparison group: Abatacept is being compared to adalimumab therapy in the trial

ELIGIBILITY:
Inclusion Criteria:

* Active rheumatoid arthritis causing pain and functional impairment with DAS28 >5.1 -Has already received usual care for inflammatory arthritis including conventional DMARD therapy e.g. methotrexate, sulfasalazine, leflunomide, hydroxychloroquine on stable dose of csDMARD for at least 4 weeks prior to study drug initiation
* Willing to participate in the study over a 12-month period
* Desirably to have positive antibodies to cyclic citrullinated peptide (ACPA/CCP)
* Between 18 and 75 years of age

Exclusion Criteria:

* Pregnancy or pregnancy planned over next 12 months
* Current or previous unsuccessful use of the biologics abatacept or adalimumab
* Co-existing other autoimmune condition, e.g. systemic lupus erythematosus, -Sjogren's syndrome, connective tissue disease, fibromyalgia, osteoarthritis, gout
* Recent surgery in the last 3 months or imminent surgery in the next 12 months
* Unable to give informed consent
* Previous history of cancer in the last 5 years
* Previous history of multiple sclerosis
* Uncontrolled heart failure, hypertension or diabetes mellitus
* Known history of fibromyalgia or other chronic pain disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Change in the Visual Analogue Score for Pain | 0, 3, 6, 9, 12 months
  The Visual Analogue Score for Pain is a pain score which has a numerical rating scale from 0 to 10
Change in the Neuropathic pain questionnaire: PainDETECT | 0, 3, 6, 9, 12 months
  The painDETECT pain questionnaire is a numerical rated score for neuropathic pain
Change in Quantitative sensory testing | 0, 3, 6, 9, 12 months
  Quantitative sensory testing measures numerical values for pain in specific regions of testing

SECONDARY OUTCOMES:
Change in Blood markers | 0, 3, 6, 9, 12 months
  Pain biomarkers in serum

CONTACTS AND LOCATIONS:
Overall Officials: Prof Sofat, MD, PhD, Principal Investigator — St George's, University of London
Locations (1):
- Hotung Centre for Musculoskeletal Diseases, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Published data will be reported in publications from the trial. Data will be shared with other researchers on written request

REFERENCES:
- [Derived] Ahmed L, Biddle K, Blundell A, Koushesh S, Kiely P, Mein G, Sedgwick P, Sofat N. Assessing the effects of distinct biologic therapies on rheumatoid arthritis pain by nociceptive, neuropathic and nociplastic pain components: a randomised feasibility study. Pilot Feasibility Stud. 2024 May 16;10(1):77. doi: 10.1186/s40814-024-01505-4. PMID 38755699